CLINICAL TRIAL: NCT05377398
Title: Effective Promotion of Healthy Lifestyles, Mental Health and Wellbeing Among Disadvantaged Groups
Brief Title: MIELITEKO Lifestyle Intervention Study
Acronym: MIELITEKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Savonia University of Applied Sciences (SAVONIA) (Unknown); City of Kuopio (Other Government); VTT Technical Research Centre of Finland (Other); Buddy Health Care (BHC) (Unknown)
Responsible Party: Principal Investigator, Tomi Mäki-Opas, Research director, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2116/02.03.01/2020
Record Dates: First submitted 2022-03-25; First posted 2022-05-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Mental Health; Well-Being; Life Style
Keywords: Mental health; Well-being; Life-style; Disadvantaged groups; intervention study; RCT; Mixed methods; Effectiveness; Registers; Digital intervention; Green power
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study is a multilayered intervention study with RCT study design. The selection of participants will be based on purposive sampling. The participants will fill in the baseline questionnaire that screens the current state of mental health, mental wellbeing and healthy lifestyle and substance use among the participants.
  Participants are then randomly allocated 1:1 to intervention (N=250) and control groups (N=250). The participants in the intervention group are offered 1) Digital individual-level intervention and 2) Individual-level or group-based intervention. In addition, all participants in the intervention group with elevated risk for substance use will also be targeted with 3) A mini-intervention for substance use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1) Intervention group (Experimental): Participants in this arm will be offered
  1. a digital individual-level intervention (Bit Habit) &
  2. group-based or individual-level healthy lifestyle and green power intervention
  3. a mini-intervention for substance use if their level of substance use is above certain risk level.
  Interventions: Behavioral: Digital individual-level intervention (Bit Habit); Behavioral: Group-based healthy lifestyle and green power intervention; Behavioral: Individual-level healthy lifestyle intervention; Behavioral: Mini-intervention for substance use
- 2) Control group (No Intervention): The control group is assumed to continue with current health information and national recommendations for healthy lifestyle and use of services "as usual".

INTERVENTIONS:
Behavioral: Digital individual-level intervention (Bit Habit) — All participants in the intervention group receive access to the BitHabit app for the 1-year intervention period. The BitHabit app was designed in the StopDia project, and it aims to help its users to adopt healthier lifestyles and habits.The content and approach of the app is based on habit formation theories and the Self-Determination Theory. The app provides an extensive library of suggested lifestyle habits that was created according to lifestyle guidelines and recommendations. The habits are related to diet, physical activity, sleep, positive mood, stress management, smoking, and alcohol consumption. Users of the app select these habits from the library to their "shopping basket" to complete in their everyday life. The app also allows the users to report and monitor their performance and progress.
  Arms: 1) Intervention group
Behavioral: Group-based healthy lifestyle and green power intervention — The group-based healthy lifestyle intervention is based on the Supportive Environment Theory (SET). The intervention is implemented in accordance with DiClemente and Prochaska's Stages-of-Change Model which is often used as framework for lifestyle change as well as Shazer and Berg's Solution Focused Brief Therapy. We expect participants to increase knowledge about healthy lifestyle choices and notice the beneficial effect of exercise, healthy diet and staying in nature. The intervention includes 12 to 16 hours of group activities during a period of 8 weeks. Interventions comprehend guided activities in nature, related to healthy relationship to food and exercise, as well as reflecting on shared experiences. In addition to group meetings, participants have access to material for mental well-being on an electronic learning environment.
  Arms: 1) Intervention group
Behavioral: Individual-level healthy lifestyle intervention — The individual-level healthy lifestyle intervention follows the principles and theoretical background of the group-based intervention, but the intervention is carried out entirely on the electronic learning environment. The participants complete activities and exercises independently or with a friend in their own time.
  Arms: 1) Intervention group
Behavioral: Mini-intervention for substance use — The mini-intervention for substance use follows the principle of the ASSIST-linked brief intervention created by WHO. This brief intervention is a phone-call lasting 3 to 15 minutes and given to the participant according to their risk score calculated with the ASSIST questionnaire which is included in the baseline survey. The intervention includes presenting the participant with their test score and associated health problems related to their level of risk. Especially in primary health care context, brief intervention according to the ASSIST score has been found to be successful in moderating risk for substance use. The intervention is not intended as a stand-alone treatment and in cases where high risk substance use is detected, the professional should encourage the participant to seek specialized drug and alcohol assessment and treatment.
  Arms: 1) Intervention group

SUMMARY:
Mental health problems cause individual, social and economic burden to the society. The mental health problems are among the highest levels in North Savo compared to the general Finnish population. The COVID-19 pandemic has emphasized the urgent need for tackling mental health problems and developing an effective and comprehensive approach to prevent mental health problems. The aim of this MIELITEKO pilot study is to test and develop an effective and comprehensive programme to prevent mental health problems and promote mental wellbeing among disadvantaged groups.

The pilot study is a multilayered intervention study with an RCT study design, which will be conducted in selected cities and areas in North Savo such as Kuopio, Iisalmi, Varkaus and Siilinjärvi. The disadvantaged groups of this study include people aged between 18 and 64 years who are unemployed or are outside the workforce. The participants are randomized 1:1 into intervention (N=250) and control groups (N=250). The intervention group will receive the multilayered intervention whereas the control group is assumed to continue with current health information and use of services "as usual" but remain in the waiting list. Multilayered intervention includes individual-level digital healthy lifestyle intervention, group-based healthy lifestyle intervention and green power intervention as well as mini-intervention for substance use.

The data collection of self-reported validated measure of health and wellbeing as well as relevant background factor will be conducted using digital and online survey tools in baseline (T0), and after 6 months (T1) and 12 months (T2) after the onset of the study from both intervention and control groups. Register data on the use of services and pharmaceuticals that will be gathered from the national registers at National Institute for Health and Welfare and Kela or from local registers administered by municipalities in North Savo. Pilot study will utilize quantitative and qualitative statistical analyses to evaluate the process, effects and effectiveness as well as cost-effectiveness of the intervention to promote mental health and wellbeing as well as to healthy lifestyles.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 64 years
* unemployed or outside the workforce (such as students)
* living in Northern Savo

Exclusion Criteria:

- no access to personal mobile devices or to the internet

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Positive Mental Health (WEMWBS) | At baseline, 6 and 12 months after baseline
  The definitive target of the healthy lifestyle intervention is an increase in measured positive mental health. The positive mental health of the respondents will be assessed with a self-reported validated measure of the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS).
  The measure consists of 14 5-point Likert scale items, where the respondent states how often during the past two weeks they have felt as described in the proposed statement (none of the time, rarely, some of the time, often, all the time). The items cover positive affect (feelings of optimism, cheerfulness, relaxation), satisfying interpersonal relationships and positive functioning (energy, clear thinking, self-acceptance, personal development, competence and autonomy). All the items are scored positively according to the Likert scale value, giving a minimum score of 14 and maximum score of 70. Higher score indicates a higher level of mental well-being.
Change in Physical Activity | At baseline, 6 and 12 months after baseline
  Physical activity is measured with assessment tools adopted from StopDia. In StopDia study, the questions regarding physical activity were modified from the Finrisk study, the Kuopio Ischaemic Heart Disease Risk Factor study and the International Physical Activity Questionnaire.
  We inquire how often and with what duration the respondents carry out planned physical activity and exercise. We also inquire with similar questions the frequency of incidental activity, for example walking the stairs or gardening. Our outcome measure of physical activity is the total time used during a week for planned or incidental conditioning and everyday physical activities.
Change in Healthy Diet Index (HDI) | At baseline, 6 and 12 months after baseline
  Diet quality and eating behaviors are assessed in the survey using the Healthy Diet Index (HDI). The Healthy Diet Index (HDI) was developed as part of the StopDia project to assess the quality of a diet. The index is a modification of the 18-Item Food Intake Questionnaire (D2D-FIQ). The index consists of seven domains: meal patterns, intake of grains, fruits and vegetables, fats, fish and meat, dairy and snacks and treats. The index is scored as a total score of the domains with a maximum score of 100 points.
Change in Alcohol, Smoking and Substance Involvement (ASSIST) | At baseline, 6 and 12 months after baseline
  Alcohol consumption, smoking and other substance use are assessed in the survey with WHO's validated ASSIST questionnaire. In the questionnaire we inquire whether the respondent has used listed substances during their lifetime or in the past three months and how often they have had a strong urge to use them. We also inquire whether the respondent has faced health, social, legal or financial difficulties because of their substance use, their friends or relatives have raised concerns or they themselves have wished to stop using the substance. The measure for alcohol, smoking and substance abuse is calculated according to the principles of the ASSIST screening tool.
Change in Pittsburgh Sleep Quality Index (PSQI) | At baseline, 6 and 12 months after baseline
  For assessment of sleep quality, we use the well-validated Pittsburgh Sleep Quality Index (PSQI). We inquire the typical times the respondent falls asleep and wakes up on weekdays and weekends. We also ask them how easy it is for them to fall asleep and if they wake up during the night. Additionally, we survey different symptoms and effects of sleep dysfunction according to the Pittsburg Sleep Quality questionnaire. Our outcome measure for sleep quality is the global PSQI score.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI 21) | At baseline, 6 and 12 months after baseline
  Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Higher score means higher depression.
Beck Anxiety Inventory (BAI 21) | At baseline, 6 and 12 months after baseline
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Higher score means higher anxiety.
Psychotic symptoms | At baseline, 6 and 12 months after baseline
  Psychotic-like experiences, Scale: Youth experiences and Health, Short version, developed by the Finnish Institute for Health and Welfare (THL), higher scores to worse to outcome.
Social inclusion scale, THL | At baseline, 6 and 12 months after baseline
  Survey instrument to assess self-reported experiences of social inclusion, summary score from individual items, scaled to 0-100, higher score means higher inclusion.
Resilience Scale (RS-14) | At baseline, 6 and 12 months after baseline
  Finnish version of the resilience scale (RS-14), shortened version of RS developed by Wagnild & Young 1993. Include 14 individual items, total score range from 14-98, higher score means higher resilience.
Capabilities (CA) | At baseline, 6 and 12 months after baseline
  Finnish versio of the capabilities scale (CA), developed by the Anand et al 2005, include 7 individual items plus summary question, scale from 1 to 7, total score is calculated by summarizing the 7 individual items, higher score means better capabilities.
UCLA loneliness scale | At baseline, 6 and 12 months after baseline
  Finnish version of the UCLA loneliness scale (Russell et al 1996), that measure Subjective feelings of loneliness as well as feelings of social isolation. Short-version, summary score in which higher scores means severe loneliness.
Social cohesion | At baseline, 6 and 12 months after baseline
  General instrument to measure trust to public institutes (government, policy, health and social care, ) and other people with a scale from 1 (low) to 5 (high trust). Summary score of these individual items presented general trust (social cohesion) to public institutes or other people. Higher score presents higher social cohesion.
The Alcohol Use Disorders Identification Test (AUDIT-C) | At baseline, 6 and 12 months after baseline
  The AUDIT-C measures whether the person's drinking is affecting his or her health and safety. Scale is scored between 0 (no use) and 12. Higher the score higher the more likely drinking is affecting health and safety of the person.
Nature relationship | At baseline, 6 and 12 months after baseline
  perceived wellbeing and health effects of the nature, including individual items on health, positive feelings, stress, importance of nature, as well as how often spends time in nature and how much per each visit. Scale for each is Likert-5, daily-once o months, not spending time - hour or more
Perceived health and illnesses | At baseline, 6 and 12 months after baseline
  persons general perception of their health and illnesses, scale (very food) 1-5 (very poor)
Diseases diagnosed by a doctor | At baseline, 6 and 12 months after baseline
  A long list of various diseases diagnosed by a doctor, scale yes or no.
Self-reported use of health and social care | At baseline, 6 and 12 months after baseline
  Use of various health and social services during the last 12 months, scale: yes or no, how many times
Register-based information of health and social service use and costs | At baseline, 6 and 12 months after baseline
  National and local register information of the use of social and health services as well as medicines will be linked to the data, including use and costs of the services and medicines

OTHER OUTCOMES:
Sociodemographic factors | At baseline, 6 and 12 months after baseline
  gender, age, marital status, education, housing, household income, size of the family, main economic activity, household income, loans, financial difficulties, reemployment possibilities

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (5):
  - University of Eastern Finland, Kuopio, Northern Savonia
  - Technical Research Centre of Finland (VTT), Espoo
  - Buddy HealthCare Ltd Oy, Helsinki
  - Savonia University of Applied Sciences (SAVONIA), Kuopio
  - City of Kuopio, Kuopio

IPD SHARING:
Plan to Share IPD: Yes
All suitable metadata produced by this study will be made openly available to the scientific community and society for example from the Finnish Social Science Data Archive (FSD). No Individual Participant Data (PDF) will be made openly available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the planned study has ended.
Access Criteria: For research purposes, persons interested to use the data can contact PI for research collaboration.

REFERENCES:
- [Background] Borodulin K, Laatikainen T, Lahti-Koski M, Jousilahti P, Lakka TA. Association of age and education with different types of leisure-time physical activity among 4437 Finnish adults. J Phys Act Health. 2008 Mar;5(2):242-51. doi: 10.1123/jpah.5.2.242. PMID 18382033
- [Background] Borodulin K, Karki A, Laatikainen T, Peltonen M, Luoto R. Daily Sedentary Time and Risk of Cardiovascular Disease: The National FINRISK 2002 Study. J Phys Act Health. 2015 Jul;12(7):904-8. doi: 10.1123/jpah.2013-0364. Epub 2014 Aug 22. PMID 25153761
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Harjumaa M, Absetz P, Ermes M, Mattila E, Mannikko R, Tilles-Tirkkonen T, Lintu N, Schwab U, Umer A, Leppanen J, Pihlajamaki J. Internet-Based Lifestyle Intervention to Prevent Type 2 Diabetes Through Healthy Habits: Design and 6-Month Usage Results of Randomized Controlled Trial. JMIR Diabetes. 2020 Aug 11;5(3):e15219. doi: 10.2196/15219. PMID 32779571
- [Background] Hemio K, Polonen A, Ahonen K, Kosola M, Viitasalo K, Lindstrom J. A simple tool for diet evaluation in primary health care: validation of a 16-item food intake questionnaire. Int J Environ Res Public Health. 2014 Mar 4;11(3):2683-97. doi: 10.3390/ijerph110302683. PMID 24599042
- [Background] Humeniuk R, Ali R, Babor T, Souza-Formigoni ML, de Lacerda RB, Ling W, McRee B, Newcombe D, Pal H, Poznyak V, Simon S, Vendetti J. A randomized controlled trial of a brief intervention for illicit drugs linked to the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) in clients recruited from primary health-care settings in four countries. Addiction. 2012 May;107(5):957-66. doi: 10.1111/j.1360-0443.2011.03740.x. Epub 2012 Feb 28. PMID 22126102
- [Background] Lakka TA, Salonen JT. Intra-person variability of various physical activity assessments in the Kuopio Ischaemic Heart Disease Risk Factor Study. Int J Epidemiol. 1992 Jun;21(3):467-72. doi: 10.1093/ije/21.3.467. PMID 1634307
- [Background] Lindstrom J, Aittola K, Polonen A, Hemio K, Ahonen K, Karhunen L, Mannikko R, Siljamaki-Ojansuu U, Tilles-Tirkkonen T, Virtanen E, Pihlajamaki J, Schwab U. Formation and Validation of the Healthy Diet Index (HDI) for Evaluation of Diet Quality in Healthcare. Int J Environ Res Public Health. 2021 Feb 28;18(5):2362. doi: 10.3390/ijerph18052362. PMID 33670967
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Pihlajamaki J, Mannikko R, Tilles-Tirkkonen T, Karhunen L, Kolehmainen M, Schwab U, Lintu N, Paananen J, Jarvenpaa R, Harjumaa M, Martikainen J, Kohl J, Poutanen K, Ermes M, Absetz P, Lindstrom J, Lakka TA; StopDia study group. Digitally supported program for type 2 diabetes risk identification and risk reduction in real-world setting: protocol for the StopDia model and randomized controlled trial. BMC Public Health. 2019 Mar 1;19(1):255. doi: 10.1186/s12889-019-6574-y. PMID 30823909
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300